CLINICAL TRIAL: NCT03353857
Title: Open-label, Randomized, Fixed Sequence Cross-over Study With Five Parallel Treatment Arms and Three Treatment Periods to Quantify the Drug-drug Interactions of Two Rifampicin Dose Strengths on Four Progestins and a Fixed Progestin-ethinylestradiol Combination Compared With Midazolam in Healthy Post-menopausal Women
Brief Title: Drug-drug Interaction Between Rifampicin and Progestins/Ethinylestradiol and Midazolam
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 19604; 2017-002792-26 (EudraCT Number)
Record Dates: First submitted 2017-11-20; First posted 2017-11-27 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Biological Availability
MeSH Terms: interventions — Levonorgestrel; Norethindrone; Desogestrel; dienogest; drospirenone; Ethinyl Estradiol; drospirenone and ethinyl estradiol combination; Midazolam; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- levonorgestrel (Experimental): levonorgestrel and midazolam will be administered on Day 1, Day 15 and Day 26. rifampicin (10 mg/day) will be administered on Day 8 to Day 18 and rifampicin (600 mg/day) on Day 19 to Day 29.
  Interventions: Drug: levonorgestrel/ Microlut; Drug: Midazolam/ Midazolam-ratiopharm; Drug: Rifampicin
- norethindrone (Experimental): norethindrone and midazolam will be administered on Day 1, Day 15 and Day 26. rifampicin (10 mg/day) will be administered on Day 8 to Day 18 and rifampicin (600 mg/day) on Day 19 to Day 29.
  Interventions: Drug: Norethindrone/ Noriday; Drug: Midazolam/ Midazolam-ratiopharm; Drug: Rifampicin
- desogestrel (Experimental): desogestrel and midazolam will be administered on Day 1, Day 15 and Day 26. rifampicin (10 mg/day) will be administered on Day 8 to Day 18 and rifampicin (600 mg/day) on Day 19 to Day 29.
  Interventions: Drug: Desogestrel/ Cerazette; Drug: Midazolam/ Midazolam-ratiopharm; Drug: Rifampicin
- dienogest (Experimental): dienogest and midazolam will be administered on Day 1, Day 15 and Day 26. rifampicin (10 mg/day) will be administered on Day 8 to Day 18 and rifampicin (600 mg/day) on Day 19 to Day 29.
  Interventions: Drug: Dienogest/ Visanne; Drug: Midazolam/ Midazolam-ratiopharm; Drug: Rifampicin
- Drospirenone/ ethinylestradiol (Experimental): drospirenone/ethinylestradiol and midazolam will be administered on Day 1, Day 15 and Day 26.
  rifampicin (10 mg/day) will be administered on Day 8 to Day 18 and rifampicin (600 mg/day) on Day 19 to Day 29.
  Interventions: Drug: Drospirenone, Ethinylestradiol/ Yasmin; Drug: Midazolam/ Midazolam-ratiopharm; Drug: Rifampicin

INTERVENTIONS:
Drug: levonorgestrel/ Microlut — In Period 1, 0.03 mg single dose administered as 1x0.03 mg tablet on Study Day 1, In Period 2, 0.03 mg single dose administered as 1x0.03 mg tablet on Study Day 15 In Period 3, 0.03 mg single dose administered as 1x0.03 mg tablet at Study Day 26
  Arms: levonorgestrel
Drug: Norethindrone/ Noriday — In Period 1, 0.35 mg single dose administered as 1x0.35 mg tablet on Study Day 1, In Period 2, 0.35 mg single dose administered as 1x0.35 mg tablet on Study Day 15 In Period 3, 0.35 mg single dose administered as 1x0.35 mg tablet at Study Day 26
  Arms: norethindrone
Drug: Desogestrel/ Cerazette — In Period 1, 0.075 mg single dose administered as 1x0.075 mg tablet on Study Day 1, In Period 2, 0.075 mg single dose administered as 1x0.075 mg tablet on Study Day 15 In Period 3, 0.075 mg single dose administered as 1x0.075 mg tablet at Study Day 26
  Arms: desogestrel
Drug: Dienogest/ Visanne — In Period 1, 2 mg single dose administered as 1x2 mg tablet on Study Day 1, In Period 2, 2 mg single dose administered as 1x2 mg tablet on Study Day 15 In Period 3, 2 mg single dose administered as 1x2 mg tablet at Study Day 26
  Arms: dienogest
Drug: Drospirenone, Ethinylestradiol/ Yasmin — In Period 1, 3 mg drospirenone, 0.03 mg ethinylestradiol single dose administered as 1x3mg drospirenone, 0.03 mg ethinylestradiol tablet on Study Day 1, In Period 2, 3 mg drospirenone, 0.03 mg ethinylestradiol single dose administered as 1x3mg drospirenone, 0.03 mg ethinylestradiol tablet on Study Day 15, In Period 3, 3 mg drospirenone, 0.03 mg ethinylestradiol single dose administered as 1x3mg drospirenone, 0.03 mg ethinylestradiol tablet on Study Day 26,
  Arms: Drospirenone/ ethinylestradiol
Drug: Midazolam/ Midazolam-ratiopharm — In Period 1, 1 mg single dose administered as 1x0.5 ml oral solution on Study Day 1, In Period 2, 1 mg single dose administered as 1x0.5 ml oral solution on Study Day 15 In Period 3, 1 mg single dose administered as 1x0.5 ml oral solution at Study Day 26
Drug: Rifampicin — In period 2, 10 mg (suspension, 0.5 ml) for 11 days at 10 mg/day In period 3, 600 mg (film-coated tablets) for 11 days at 600 mg/day

SUMMARY:
Quantify the effect of a probe CYP3A4 inducer (Rifampicin) on the pharmacokinetics of levonorgestrel, norethindrone, desogestrel, dienogest, drospirenone,estradiol and midazolam

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subject based on a complete medical history, physical examination, ECG, and clinical laboratory tests
* Age: 45 to 70 years (inclusive) at the first screening visit
* Minimum body weight 50 kg with Body mass index (BMI) above or equal to 18.5 kg/m², and below or equal to 30 kg/m² at the first screening visit
* Postmenopausal state, revealed indicated by either:

  * medical history, if applicable (natural menopause at least 12 months prior to first study drug administration, for women younger than 60 years confirmed by follicle stimulating hormone (FSH) >40 IU/L AND estradiol ≤ 20 pg/mL; or
  * surgical menopause by bilateral ovariectomy at least 3 months prior to first study drug administration)

Exclusion Criteria:

* Relevant diseases within the last 4 weeks prior to the first study drug administration, i.e. any disease requiring treatment by a health-care provider
* Febrile illness within 1 week before the first study drug administration
* Known severe allergies, non-allergic drug reactions, or multiple drug allergies
* Presence or history of thrombosis, thrombophlebitis, thromboembolic diseases of veins and/or arteries, e.g. deep vein thrombosis, stroke, myocardial infarction, pulmonary embolism, transient ischemic attack, angina pectoris
* Presence or history of conditions that increase the risk of thromboembolic diseases, e.g. disturbances of the coagulation system, thromboembolic diseases in close relatives at age ≤50 years], valvular heart disease, atrial fibrillation, cardiac dysfunction)
* Presence, history, or suspected presence of malignant tumors or tumors of the liver and pituitary
* Presence or history of liver disease e.g. disturbances of the bilirubin excretion (Dubin-Johnson and Rotor syndromes), cholecystectomy ; cholestasis, idiopathic icterus or pruritus during a previous pregnancy or estrogen-progestogen treatment
* Relevant kidney diseases or renal injury associated with multisystem diseases/disorders, e.g. glomerulonephritis systemic lupus erythematous, diabetic nephropathy. A history of a single episode of uncomplicated nephrolithiasis does not prevent participation
* Known metabolic disorder, e.g. diabetes mellitus, severe hypertriglyceridemia
* Migraine with neurologic symptoms
* Clinically significant depression, current or in the last year
* Known current thyroid disorders which require treatment. Subjects with an euthyroid struma who do not need any treatment can participate.
* Chronic respiratory insufficiency
* History of porphyria
* Contraindications for midazolam, e.g. myasthenia gravis, and sleep apnea

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2018-07-04 (Actual); Study Completion 2019-02-19 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration time curve from zero to infinity (AUC) of levonorgestrel in the presence of MDZ (without RIF) and in combination with 10 mg/d and 600 mg/d RIF | Over 7 days in Period 1 (no RIF) and 4 days in treatment Periods 2 and 3
Maximum plasma concentration (Cmax) of levonorgestrel in the presence of MDZ (without RIF) and in combination with 10 mg/d and 600 mg/d RIF | Over 7 days in Period 1 (no RIF) and 4 days in treatment Periods 2 and 3
Area under the plasma concentration time curve from zero to infinity (AUC) of norethindrone in the presence of MDZ (without RIF) and in combination with 10 mg/d and 600 mg/d RIF | Over 7 days in Period 1 (no RIF) and 4 days in treatment Periods 2 and 3
Maximum plasma concentration (Cmax) of norethindrone in the presence of MDZ (without RIF) and in combination with 10 mg/d and 600 mg/d RIF | Over 7 days in Period 1 (no RIF) and 4 days in treatment Periods 2 and 3
Area under the plasma concentration time curve from zero to infinity (AUC) of etonogestrel in the presence of MDZ (without RIF) and in combination with 10 mg/d and 600 mg/d RIF | Over 7 days in Period 1 (no RIF) and 4 days in treatment Periods 2 and 3
Maximum plasma concentration (Cmax) of etonogestrel in the presence of MDZ (without RIF) and in combination with 10 mg/d and 600 mg/d RIF | Over 7 days in Period 1 (no RIF) and 4 days in treatment Periods 2 and 3
Area under the plasma concentration time curve from zero to infinity (AUC) of dienogest in the presence of MDZ (without RIF) and in combination with 10 mg/d and 600 mg/d RIF | Over 7 days in Period 1 (no RIF) and 4 days in treatment Periods 2 and 3
Maximum plasma concentration (Cmax) of dienogest in the presence of MDZ (without RIF) and in combination with 10 mg/d and 600 mg/d RIF | Over 7 days in Period 1 (no RIF) and 4 days in treatment Periods 2 and 3
Area under the plasma concentration time curve from zero to infinity (AUC) of drospirenone (+EE) in the presence of MDZ (without RIF) and in combination with 10 mg/d and 600 mg/d RIF | Over 7 days in Period 1 (no RIF) and 4 days in treatment Periods 2 and 3
Maximum plasma concentration (Cmax) of drospirenone (+EE) in the presence of MDZ (without RIF) and in combination with 10 mg/d and 600 mg/d RIF | Over 7 days in Period 1 (no RIF) and 4 days in treatment Periods 2 and 3
Area under the plasma concentration time curve from zero to infinity (AUC) of ethinylestradiol (+DRSP) in the presence of MDZ (without RIF) and in combination with 10 mg/d and 600 mg/d RIF | Over 7 days in Period 1 (no RIF) and 4 days in treatment Periods 2 and 3
Maximum plasma concentration (Cmax) of ethinylestradiol (+DRSP) in the presence of MDZ (without RIF) and in combination with 10 mg/d and 600 mg/d RIF | Over 7 days in Period 1 (no RIF) and 4 days in treatment Periods 2 and 3
Area under the plasma concentration time curve from zero to infinity (AUC) of midazolam in combination with the hormonal contraceptive only (without RIF) and in combination with 10 mg/d and 600 mg/d RIF | Over 7 days in Period 1 (no RIF) and 4 days in treatment Periods 2 and 3
Maximum plasma concentration (Cmax) of midazolam in combination with the hormonal contraceptive only (without RIF) and in combination with 10 mg/d and 600 mg/d RIF | Over 7 days in Period 1 (no RIF) and 4 days in treatment Periods 2 and 3

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - CRS Clinical-Research-Services Mannheim GmbH, Mannheim, Baden-Wurttemberg
  - CRS Clinical-Research-Services Mönchengladbach GmbH, Mönchengladbach, North Rhine-Westphalia

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/